CLINICAL TRIAL: NCT00199849
Title: Safety and Immunological Evaluation of NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine Given by Particle-mediated Epidermal Delivery (PMED) in Patients With Tumor Type Known to Express NY-ESO-1 or LAGE-1 Antigen.
Brief Title: NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: New York Presbyterian Hospital (Other); M.D. Anderson Cancer Center (Other); Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0013; LUD2002-006 (Other: Ludwig Institute for Cancer Research)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2021-10-08 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer; Bladder Cancer; Non-small Cell Lung Cancer; Esophageal Cancer; Sarcoma
Keywords: NY-ESO-1; DNA
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (3):
- Cohort 1 (Experimental): 4 µg NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine
  NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered by particle-mediated epidermal delivery (PMED) at a pressure of 500 psi using the XR-1 Powderject® delivery device. The 4 µg dosage of NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered as 4 X 1 µg PMEDs in close proximity.
  The vaccine was administered in weeks 1, 5, and 9 of Cycle 1. In the absence of > Grade 3 toxicity and in the absence of progressive disease requiring other treatment or the presence of NY-ESO-1 immunity, patients could receive an additional cycle of vaccinations of NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine.
  Interventions: Biological: NY-ESO-1 Plasmid DNA Cancer Vaccine
- Cohort 2 (Experimental): 8 µg NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine
  NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered by particle-mediated epidermal delivery (PMED) at a pressure of 500 psi using the XR-1 Powderject® delivery device.
  The 8 µg dosage of NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered as 8 X 1 µg PMEDs.
  The vaccine was administered in weeks 1, 5, and 9 of Cycle 1. In the absence of > Grade 3 toxicity and in the absence of progressive disease requiring other treatment or the presence of NY-ESO-1 immunity, patients could receive an additional cycle of vaccinations of NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine.
  Interventions: Biological: NY-ESO-1 Plasmid DNA Cancer Vaccine
- Cohort 3 (Experimental): 8 µg NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine
  NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered by particle-mediated epidermal delivery (PMED) at a pressure of 500 psi using the XR-1 Powderject® delivery device.
  The 8 µg dosage of NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered as a cluster dosage of 4 doses (day 1, 3, 5, 8) as 2 X 1 µg PMEDs per day.
  The vaccine was administered in weeks 1, 5, and 9 of Cycle 1. In the absence of > grade 3 toxicity and in the absence of progressive disease requiring other treatment or the presence of NY-ESO-1 immunity, patients could receive an additional cycle of vaccinations of NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine.
  Interventions: Biological: NY-ESO-1 Plasmid DNA Cancer Vaccine

INTERVENTIONS:
Biological: NY-ESO-1 Plasmid DNA Cancer Vaccine — NY-ESO-1 Plasmid DNA Cancer Vaccine administered by particle-mediated epidermal delivery (PMED) at a pressure of 500 psi using the XR-1 Powderject® delivery device.

SUMMARY:
To evaluate the safety of NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine given by particle-mediated epidermal delivery (PMED) in patients with tumor types known to express NY-ESO-1 or LAGE-1.

DETAILED DESCRIPTION:
NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered by particle-mediated epidermal delivery (PMED) at a pressure of 500 psi using the XR-1 Powderject® delivery device. The 4 microgram dosage of NY-ESO-1 was administered as 4 X 1 microgram PMEDs in close proximity. Similarly, the 8 microgram dosage was administered as 8 X 1 microgram PMEDs. The third cohort of patients received the 8 microgram dosage as a cluster dosage of 4 doses (day 1, 3, 5, 8) as 2 X 1 microgram PMEDs per day.

Blood samples were to be obtained at baseline, 2 weeks after each vaccination, prior to the second and third vaccination, and 4 weeks after the third vaccination for the assessment of clinical hematology, biochemistry measurements and immunology responses. Patients were to be evaluated for toxicity throughout the study.

Delayed-type hypersensitivity (DTH) testing was to be performed at baseline and at the 2-week visit following the first and third vaccinations.

NY-ESO-1 and/or LAGE-1 specific antibodies were to be assessed in all patients by an enzyme-linked immunosorbent assay (ELISA). NY-ESO-1 specific CD4+ and CD8+ T-cells were to be assessed in all patients by tetramer and/or ELISPOT assays.

Disease status was to be assessed at baseline and 4 weeks after the third vaccination in patients with measurable disease.

ELIGIBILITY:
Inclusion Criteria:

Patients were eligible for enrollment if they fulfilled all of the following criteria:

1. Histologically proven tumor type known to express NY-ESO-1 or LAGE-1 (prostate cancer, breast cancer, bladder cancer, hepatocellular cancer, synovial sarcoma, leiomyosarcoma, head and neck, lung cancer, esophageal, ovarian, neuroblastoma); or NY-ESO-1 or LAGE-1 positive tumors determined by reverse transcriptase and polymerase chain reaction (RT-PCR) analysis, preferably, or immunohistochemistry or expression of LAGE-1 by RT-PCR.
2. Advanced disease and have declined, delayed, failed or completed standard therapy.
3. Full recovery from surgery.
4. Expected survival of at least 6 months.
5. Karnofsky performance scale ≥ 60.
6. Adequate bone marrow, kidney, liver and immune functions.
7. Able and willing to give valid written informed consent.

Exclusion Criteria:

1. Clinically significant heart disease (NYHA Class III or IV).
2. Other serious illnesses, e.g., serious infections requiring antibiotics or bleeding disorders, clinically significant liver or renal insufficiency requiring treatment.
3. Patients with serious intercurrent illness, requiring hospitalization.
4. Known HIV, Hepatitis B or Hepatitis C positivity.
5. History of autoimmune diseases (e.g. SLE, scleroderma). Vitiligo is not an exclusion criterion.
6. Concomitant systemic treatment with corticosteroids, anti-histaminic drugs or non-steroidal anti-inflammatory drugs. Specific COX-2 inhibitors are permitted. Low dose aspirin is permitted. Topical or inhalational steroids are permitted.
7. Evidence of skin disease (e.g. psoriasis, eczema or keloid formation) at the proposed administration site.
8. Allergy to gold (including gold jewelry).
9. History or evidence of chrysotherapy (gold salts).
10. Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to first dosing (6 weeks for nitrosoureas).
11. Other malignancy within 3 years prior to entry into the study, except for treated non-melanoma skin cancer, cervical carcinoma in situ.
12. Mental impairment, in the opinion of the investigator, that may compromise the ability to give informed consent and comply with the requirements of the study.
13. Lack of availability for immunological and clinical follow-up assessments.
14. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dosing.
15. Pregnancy or breastfeeding.
16. Women of childbearing potential: Refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-09-27 (Actual); Primary Completion 2006-09-11 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Padmanee Sharma, MD PhD, Principal Investigator — UT MD Anderson Cancer Center Genitourinary Med Onc; Nasser K Altorki, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - New York Presbyterian Hospital, New York, New York
  - UT MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 4 µg NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine
  NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered by particle-mediated epidermal delivery (PMED) at a pressure of 500 psi using the XR-1 Powderject® delivery device.
  The 4 µg dosage of Plasmid DNA (pPJV7611) Cancer Vaccine was administered as 4 X 1 µg PMEDs in close proximity.
  The vaccine was administered in weeks 1, 5, and 9.
- Cohort 2: 8 µg NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine
  NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered by particle-mediated epidermal delivery (PMED) at a pressure of 500 psi using the XR-1 Powderject® delivery device.
  The 8 µg dosage of NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered as 8 X 1 µg PMEDs.
  The vaccine was administered in weeks 1, 5, and 9.
- Cohort 3: 8 µg NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine
  NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered by particle-mediated epidermal delivery (PMED) at a pressure of 500 psi using the XR-1 Powderject® delivery device.
  The 8 µg dosage of NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered as a cluster dosage of 4 doses (day 1, 3, 5, 8) as 2 X 1 µg PMEDs per day.
  The vaccine was administered in weeks 1, 5, and 9.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 3 | 7 | 8
Completed | 3 | 6 | 6
Not Completed | 0 | 1 | 2
Not completed — Unrelated illness or complication | 0 | 1 | 0
Not completed — Progressive disease requiring intervention | 0 | 0 | 1
Not completed — Did not meet eligibility criteria - not dosed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of NY-ESO-1 Plasmid DNA Vaccine.
Groups:
- Cohort 1: 4 µg NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine
  NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered by particle-mediated epidermal delivery (PMED) at a pressure of 500 psi using the XR-1 Powderject® delivery device.
  The 4 µg dosage of NY-ESO-1 Plasmid DNA (pPJV7611) Cancer Vaccine was administered as 4 X 1 µg PMEDs.
  The vaccine was administered in weeks 1, 5, and 9.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 3 | 7 | 7 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5 | 10
  >=65 years | 1 | 4 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 2
  Male | 1 | 7 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 7 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 7 | 7 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicities (DLTs) and Number of Patients With Adverse Events
Description: All adverse events were graded according to the National Cancer Institute Common Toxicity Criteria (CTC) Scale (Version 3.0, published June 10, 2003).
  DLT was defined as
  * ≥ Grade 2 autoimmune phenomena
  * Asymptomatic bronchospasm or generalized urticaria
  * Grade ≥ non hematological toxicities (including injection site reactions)
  * Grade ≥ 3 hematological toxicities
  A dose-limiting adverse event must be definitely, probably, or possibly related to the administration of the investigational agent and must occur between first dose and 4 weeks after the last dose.
Time Frame: up to 13 weeks
Population: All patients who received at least one dose of NY-ESO-1 Plasmid DNA Vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 7 | 7
Participants
  Number of patients with DLTs | 0 | 0 | 0
  Number of patients reporting adverse events | 3 | 7 | 7

2. Secondary Outcome: Number of Patients With Tumor Response According to the Response Evaluation Criteria in Solid Tumors (RECIST).
Description: Tumor response was assessed in patients with measurable tumors according to the Response Evaluation Criteria in Solid Tumors (RECIST).
  Computed tomography (CT) scans were performed at screening and at week 13. Response was assessed using RECIST version 1.0 (Therasse et al, J Natl Cancer Inst 2000; 92:205-16). Per RECIST, target lesions are categorized as follows: complete response (CR): disappearance of all target lesions (no evaluable disease); partial response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; stable disease (SD): small changes that do not meet above criteria; no evidence of disease (NED): no new lesions in patients who did not have target lesions at baseline.
Time Frame: 13 weeks
Population: All patients who received at least one dose of NY-ESO-1 Plasmid DNA Vaccine and had valid tumor response measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 6 | 7
Participants
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0
  Stable Disease (SD) | 2 | 1 | 2
  Progressive Disease (PD) | 1 | 2 | 5
  No Evidence of Disease (NED) | 0 | 3 | 0

3. Secondary Outcome: Number of Patients With NY-ESO-1-Specific Humoral Immunity as Determined by an Increase in Antibody Titer From Baseline.
Description: Blood samples were obtained at baseline (prior to the first dose), and in weeks 3, 5, 7, 9, 11 and 13 for the assessment of NY-ESO-1-specific antibodies by an enzyme-linked immunosorbent assay (ELISA). A positive response was a readable optical density at 280 nm.
Time Frame: up to 13 weeks
Population: All patients who received at least one dose of NY-ESO-1 Plasmid DNA Vaccine and had baseline and at least one post-treatment sample taken. One patient in Cohort 3 did not have a baseline sample taken.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 7 | 6
Participants
  Number of patients with negative titers both pre-and post-treatment | 3 | 7 | 6
  Number of patients with negative titers at baseline and positive titers after treatment | 0 | 0 | 0

4. Secondary Outcome: Number of Patients With NY-ESO-1-Specific Cellular Immunity as Measured by an Increase in NY-ESO-1-Specific CD4+ and CD8+ T-Cells Following Treatment.
Description: Blood samples were obtained at baseline (prior to the first dose), and in weeks 3, 5, 7, 9, 11 and 13 for the assessment of NY-ESO-1-specific CD4+ and CD8+ T-cell responses by ELISPOT.
Time Frame: up to 13 weeks
Population: All patients who received at least one dose of NY-ESO-1 Plasmid DNA Vaccine and had baseline and at least one post-treatment sample taken. One patient in Cohort 2 did not have samples taken. All patients did not have samples analyzed for CD8+ T-cell responses.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 6 | 7
Participants
  Number of patients with an increase in CD4+ T-cells | 3 | 5 | 7
  Number of patients without an increase in CD4+ T-cells | 0 | 1 | 0
  Number of patients with an increase in CD8+ T-cells: number analyzed (Participants) | 3 | 4 | 4
  Number of patients with an increase in CD8+ T-cells | 1 | 0 | 1
  Number of patients without an increase in CD8+ T-cells: number analyzed (Participants) | 3 | 4 | 7
  Number of patients without an increase in CD8+ T-cells | 2 | 4 | 4

5. Secondary Outcome: Number of Patients With Delayed-Type Hypersensitivity (DTH) Skin Reactions to NY-ESO-1 Protein
Description: Delayed-Type Hypersensitivity (DTH) testing was conducted at baseline and on days 15 and 72 of the study. A positive DTH reaction to NY-ESO-1 protein at baseline was absent in all patients. The presence of redness and induration was considered necessary for a positive DTH reaction.
Time Frame: Up to 11 weeks
Population: All patients who received at least one dose of NY-ESO-1 Plasmid DNA Vaccine and had baseline and at least one post-treatment sample taken.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 3 | 7 | 7
Participants
  Number of Patients With DTH Skin Reactions | 0 | 3 | 1
  Number of Patients Without DTH Skin Reactions | 3 | 4 | 6

ADVERSE EVENTS:
Time Frame: up to 13 weeks
Description: All Adverse Events (AEs) were to be documented in the source records and on the respective Case Report Form (CRF) pages. Events, which occurred after signed informed consent, but before first administration of study medication, were to be documented on the Pre-existing Signs and Symptoms CRF page. Thereafter, they were documented on the Adverse Event pages. AEs were graded according to the National Cancer Institute Common Toxicity Criteria (CTC) Scale (Version 3.0, published June 10, 2003).
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/7 | 1/7
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=7) | Cohort 3 (N=7)
Pyrexia (General disorders) | 1 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 1 | 0
Hemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=7) | Cohort 3 (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Anthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Aspartate transaminase increased (Investigations) | 0 | 0 | 1
Bilirubin increased (Investigations) | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 2
Blood urea increased (Investigations) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Chest pain (Cardiac disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Dizziness (Vascular disorders) | 0 | 1 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 3 | 4
Headache (Nervous system disorders) | 1 | 1 | 3
Hematuria (Renal and urinary disorders) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Hot flush (General disorders) | 0 | 0 | 1
Hyperglycemia (Endocrine disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2
Hypoglycemia (Endocrine disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0
Injection site reaction (General disorders) | 3 | 7 | 7
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Mood alteration (Psychiatric disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 1
Peripheral edema (Cardiac disorders) | 0 | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No